CLINICAL TRIAL: NCT00560781
Title: Targeting Cognition in PTSD: Pregnenolone Augmentation of SSRIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VA IRB# 01023
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Pregnenolone; Cognition
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Pregnenolone
  Interventions: Drug: Pregnenolone or Placebo
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Pregnenolone or Placebo

INTERVENTIONS:
Drug: Pregnenolone or Placebo — Pregnenolone 50 mg BID, Pregnenolone 150 mg BID, Pregnenolone 250 mg BID

SUMMARY:
This study will test the therapeutic potential of augmenting a stable SSRI regimen with the neurosteroid pregnenolone to reduce cognitive symptoms and PTSD symptoms in patients diagnosed with PTSD.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age, any ethnic group, either sex
2. DSM-IV diagnosis of PTSD by MINI (see schedule of events)
3. No change in SSRI medications for > 4 weeks.
4. No anticipated need to alter any psychotropic medications for the 10-week duration of the study.
5. Ability to fully participate in the informed consent process, or have a legal guardian able to participate in the informed consent process.

Exclusion Criteria:

1. Unstable medical or neurological illness, including seizures, CVA, prostate or breast cancer
2. Use of oral contraceptives or other hormonal supplementation such as estrogen.
3. Significant suicidal or homicidal ideation.
4. Concomitant medications for medical conditions will be addressed on a case-by-case base to determine if exclusionary.
5. Current DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition; history of substance dependence within the last 3 months
6. Female patients who are pregnant or breast-feeding.
7. Known allergy to study medication.
8. Drugs with a narrow therapeutic index (e.g. thioridazine, mesoridazine, ziprasidone, clozapine, etc.) will be excluded, as suggested by the FDA; patients taking these agents will not be eligible for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
CAPS, BAC-A | Prospective

SECONDARY OUTCOMES:
PCL, CD-RISC, CGI, BDI-II | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD MA, Principal Investigator — Durham VAMC
Locations (1):
- Durham VAMC, Durham, North Carolina, United States